CLINICAL TRIAL: NCT02901340
Title: Third Trimester Fetal Renal Artery Doppler Indices in Borderline Idiopathic Isolated Oligohydramnios and Relationship Between Neonatal Outcomes
Brief Title: Fetal Renal Artery Doppler Indices in Borderline Isolated Oligohydramnios
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erdem Sahin, Principal Investigator, Kayseri Education and Research Hospital
Other Study IDs: 2016/474
Record Dates: First submitted 2016-09-04; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Oligohydramnios
Keywords: Borderline idiopathic isolated oligohydramnios; Fetal renal artery doppler indices; neonatal outcomes; Maternal hydration
MeSH Terms: conditions — Oligohydramnios

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Borderline isolated oligohydramnios: Borderline idiopathic isolated oligohydramnios was defined according to the four quadrants technical with ultrasound examination and diagnosed with amniotic fluid index>5.0 and ≤8.0cm.
  The borderline idiopathic isolated oligohydramnios group was formed of the patients who meets the inclusion criteria and between 34-37 weeks gestation (n:40)
  Interventions: Dietary Supplement: one to two liters of water daily
- Control group: The control group was formed of the patients who had normal amniotic volume and 34-37 weeks gestation who meets the inclusion criteria (n:100)

INTERVENTIONS:
Dietary Supplement: one to two liters of water daily
  Groups: Borderline isolated oligohydramnios

SUMMARY:
The purpose of the study is to investigate third trimester fetal renal artery doppler indices in borderline idiopathic isolated oligohydramnios and relationship between neonatal outcomes.

DETAILED DESCRIPTION:
During a routine pregnancy examination at 34-37 weeks gestation, the fetus was evaluated using ultrasound with the Toshiba Xario 200 3.5-megahertz probe. Fetal biometric measurements were obtained and placental structure and the amniotic fluid amount were evaluated in four quadrants. After detailed ultrasonography of the fetus, eligible pregnant women were included in the study.

Borderline idiopathic isolated oligohydramnios was defined according to the four quadrants technical with ultrasound examination and diagnosed with amniotic fluid index >5.0 and ≤8.0cm. After first ultrasound examination all patients in borderline isolated oligohydramnios group were hydrated with one to two liters of water daily. All patients monitored with non stress test and amniotic fluid index twice weekly until delivery after treatment with hydration.

For evaluating renal artery blood flow, an axial image of the fetal abdomen was obtained at the level of the fetal kidneys. Using color flow Doppler, the renal arteries were evaluated at the level of their origin from the abdominal aorta. The Doppler gate was placed within the lumen in a straight segment of the vessel. A minimum of three consecutive waveforms was used to calculate the PI. The umbilical artery Doppler measurements were studied in a free loop of cord, far from the fetus and placenta. pulsatile index and resistance index values were recorded.

The study consisted of two groups. The first group was formed of the patients who had normal amniotic volume and meets the inclusion criteria. In second group the investigators included patients who diagnosed borderline idiopathic isolated oligohydramnios. After delivery the investigators compared fetal renal artery doppler indices and neonatal outcomes between groups.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancies
* between 34-37 gestational weeks
* the age of them ranged from 18 to 35 years

Exclusion Criteria:

* uteroplacental insufficiency
* preeclampsia
* chronic hypertension
* collagen vascular disease
* nephropathy
* chromosomal abnormalities
* congenital abnormalities, especially those associated with impaired urine production
* growth restriction
* ruptured fetal membranes
* twin pregnancies

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population was consisted of 2 groups and included pregnant women in between 34 and 37. weeks of gestation for both groups. The normal pregnancy group was consisted of 100 healthy pregnant women whom excluded borderline idiopathic isolated oligohydramniosis , the main group was consisted of 40 pregnant women with diagnosed borderline idiopathic isolated oligohydramniosis.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Fetal renal artery pulsatile index in borderline idiopathic isolated oligohydramnios | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri Training and Research Hospital, Kayseri, Turkey (Türkiye)